CLINICAL TRIAL: NCT03607955
Title: Phase IB Study of Paclitaxel + Carboplatin With AVB-S6-500 in Women With Stage III or IV Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer Receiving Neoadjuvant Chemotherapy
Brief Title: Paclitaxel + Carboplatin With AVB-S6-500 in Women With Stage III or IV Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer Receiving Neoadjuvant Chemotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial may move forward as an NCI-sponsored trial and not an investigator initiated trial.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-x211
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AVB-S6-500 + Paclitaxel + Carboplatin (Experimental): * Paclitaxel will be given intravenously at a dose of 175 mg/m^2 on an outpatient basis over 3 hours on Day 1 of each 21-day cycle
  * Carboplatin will be given intravenously at a dose of AUC 6 over 30 minutes on Day 1 of each cycle of chemotherapy
  * AVB-S6-500 will be given at doses based on the dose escalation schema
  * The investigators will continue dosing AVB-S6-500 until 1 week prior to surgery and continuing after surgery. Maintenance dosing q2 weeks will begin with Cycle 7A/7B and be given every 2 weeks for 12 months through Cycle 19 (total of 13 maintenance cycles).
  Interventions: Drug: AVB-S6-500; Drug: Paclitaxel; Drug: Carboplatin; Procedure: Tissue from Diagnostic Laparoscopy; Procedure: Tissue from Core biopsy; Procedure: Interval Debulking; Procedure: Peripheral blood; Procedure: Ascites collection

INTERVENTIONS:
Drug: AVB-S6-500 — AVB-S6-500 is supplied by Aravive Biologics
Drug: Paclitaxel — Commercially available
  Other Names: Taxol
Drug: Carboplatin — Commercially available
  Other Names: Paraplatin
Procedure: Tissue from Diagnostic Laparoscopy — -For patients scheduled to undergo a diagnostic laparoscopy for tissue diagnosis prior to neoadjuvant chemotherapy, a tissue biopsy section from the ovary or an intra-abdominal implant will be performed
Procedure: Tissue from Core biopsy — -Standard of care procedure but research specimens will be collected
Procedure: Interval Debulking — * Standard of Care
  * Research tissue samples will be collected
Procedure: Peripheral blood — -Before initiation of neoadjuvant chemotherapy and at the time of interval debulking surgery either pre-operatively, intraoperatively, or post-operatively.
Procedure: Ascites collection — -A total of 25-100ml of ascites will be collected prior to chemotherapy treatment, if available.

SUMMARY:
The receptor tyrosine kinase AXL is a pathway that plays a crucial role in metastasis and chemoresistance. Overexpression of AXL has been associated with metastasis, recurrence, and chemoresistance in various cancer including ovarian cancer[16, 17]}. Targeting AXL is an attractive approach because it is overexpressed among patients with epithelial ovarian cancer and strongly associated with advanced stages, high grade cancer and shorter median survival time. AVB-S6-500 is a potent AXL inhibitor by binding to the ligand Gas6. Pre-clinical studies found that AVB-S6-500 was efficacious in ovarian cancer xenograft tumor models. Interventions which would increase the proportion of patients achieving pCR in this patient population could impact survival favorably and are of interest for study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal cancer per pre-treatment biopsies by laparoscopy or interventional radiology or CT-guided core biopsy.
* Patients with the following histologic epithelial cell types are eligible:

  * High grade serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelia carcinoma
  * Adenocarcinoma not otherwise specified (NOS)
* Disease must be considered "bulky" by the clinician (unresectable via primary debulking surgery) and in need of neoadjuvant chemotherapy prior to debulking surgery. This assessment of unresectability can be made via imaging or laparoscopic scoring.
* Must have pre-treatment tumor tissue available or agree to tissue collection from IR-guided biopsy.
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (unless liver metastases are present in which case AST/ALT must be ≤ 5.0 x IULN)
  * Serum creatinine < 2.0 mg/dL or < 177 µmol/L OR calculated or measured creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault equation)
  * INR ≤ 1.5 x IULN
  * aPTT ≤ 1.5 x IULN
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Any prior treatment with AVB-S6-500 or standard of care drugs (cisplatin, carboplatin, paclitaxel).
* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only. Patients with concomitant endometrial cancer diagnosed at the time of the ovarian cancer are allowed to participate if the endometrial cancer is FIGO stage IB or less.
* Currently receiving any other (non-study) cytotoxic chemotherapy.
* Currently receiving any other investigational agents or has received an investigational agent within 4 weeks of start of study treatment.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to AVB-S6-500 or other agents used in the study.
* Abnormal gastrointestinal function (nausea or vomiting). This includes GI obstruction or bleeding or signs/symptoms thereof within 3 months of study enrollment. Patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula.
* Significant cardiac disease history including:

  * Clinically significant atrial or ventricular arrhythmias requiring treatment
  * Medically controlled congestive heart failure
  * Significant angina or clinically and/or electrocardiographically documented myocardial infarction within the past year
  * Clinically significant valvular disease
* Non-healing wound, ulcer, or bone fracture.
* Receiving treatment for active autoimmune disease. "Active" refers to any condition currently requiring therapy.
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration and the patient remains free of recurrent or metastatic disease.
* Received prior chemotherapy for any abdominal or pelvic tumor. Prior adjuvant chemotherapy for localized breast cancer is permitted, provided that was completed more than 3 years prior to registration and the patient remains free of recurrent or metastatic disease.
* Known active hepatitis; ongoing systemic bacterial, fungal, or viral infection; known HIV infection or AIDS-related illness.
* History or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, or history of CVA, TIA, or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* History of major surgical procedure within 21 days prior to start of study treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | Completion of the enrollment and treatment of all patients (estimated to be approximately 26 months)
  * The study will employ the Bayesian optimal interval design (BOIN) to find the MTD.
  * Select as the MTD the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there are ties, select the higher dose level when the isotonic estimate is lower than the target toxicity rate and select the lower dose level when the isotonic estimate is greater than or equal to the target toxicity rate.
Dose limiting toxicities (DLTs) of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | Through completion of 1st cycle for all patients (estimated to be 13 months)
  -Hematologic DLT any of the following that occur during the 1st cycle (C) that are possibly (pos), probably (prob), or definitely (def) related to the study treatment:
  * Grade (Gr.) 4 neutropenia or thrombocytopenia > 7 day
  * Febrile neutropenia w/ temp > 38.5 °C
  * Gr. 4 anemia or Gr. 4 thrombocytopenia which requires transfusion therapy on more than 2 occasions in 7 days
  * Gr. thrombocytopenia w/ bleeding
  Non-hematologic DLT is any pos, prob, or def related Gr. 3 or grade 4 non-hematologic toxicity that occurs during C1 with the following exceptions:
  * Gr. 3/4 nausea/vomiting/anorexia that returns to Gr. 1 prior to the start of C2
  * Gr. 3 nausea/vomiting or diarrhea < 72 hours with adequate antiemetic and other supportive care starting with C2
  * Gr. 3 triglycerides will only be considered a DLT for patients who have grade 3 in spite of appropriate lipid lowering drug therapy
  * Gr. 3 rash (patients who have received 2 weeks of supportive care treatment w/ no improvement)
Tolerability of the combination at the MTD of AVB-S6-500 assessed in combination with standard neoadjuvant chemotherapy as measured by treatment discontinuation | Through completion of treatment (estimated to be 14 months)
Tolerability of the combination at the MTD of AVB-S6-500 assessed in combination with standard neoadjuvant chemotherapy as measured by number of dose interruption/reductions | Through completion of treatment (estimated to be 14 months)
Tolerability of the combination at the MTD of AVB-S6-500 assessed in combination with standard neoadjuvant chemotherapy as measured by use of supportive therapies | Through completion of treatment (estimated to be 14 months)
Tolerability of the combination at the MTD of AVB-S6-500 assessed in combination with standard neoadjuvant chemotherapy as measured by number of hospital admissions | Through completion of treatment (estimated to be 14 months)
Tolerability of the combination at the MTD of AVB-S6-500 assessed in combination with standard neoadjuvant chemotherapy as measured by number of deaths | Through completion of treatment (estimated to be 14 months)

SECONDARY OUTCOMES:
Objective clinical response (cOR) of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | At the time of interval debulking (approximately 9-12 weeks)
  -cOR = clinical response seen at the time of surgery with no visible disease
Pathological complete response (pCR) at the time of interval debulking surgery of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | At the time of interval debulking (approximately 9-12 weeks)
  -pCR = pathological response seen by the pathology at the time of surgery with treatment effect and no disease seen microscopically
Progression-free survival (PFS) at 1 year after debulking surgery of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | 1 year after debulking surgery (approximately 64 weeks)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Progression-free survival (PFS) at 2 years after debulking surgery of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | 2 years after debulking surgery (approximately 116 weeks)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Overall survival (OS) by long-term follow-up of AVB-S6-500 in combination with and following conventional chemotherapy and maintenance | 5 years after completion of treatment (approximately 74 months)
  -OS is defined as the time from the date of treatment to the date of death, censored at the last follow-up otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Fuh, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu